CLINICAL TRIAL: NCT05562882
Title: A Investigator-initiated Clinical Trial to Assess Safety and Efficacy of Daratumumab in the Treatment of Relapsed/Refractory Primary Immune Thrombocytopenia
Brief Title: A Clinical Trial to Assess Safety and Efficacy of Daratumumab in the Treatment of Primary Immune Thrombocytopenia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2022039（1）; 2022-D-ITP (Other: CAMS&PUMC)
Record Dates: First submitted 2022-09-28; First posted 2022-10-03 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2024-05

CONDITIONS: Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — daratumumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Daratumumab once a week x 8 doses
  Interventions: Drug: Daratumumab Injection

INTERVENTIONS:
Drug: Daratumumab Injection — intravenous daratumumab administration
  Other Names: Darzalex

SUMMARY:
A single-center, open-label, off-label use investigator-initiated clinical study to explore the clinical activity and safety of daratumumab in adult ITP patients who have not responded adequately or relapsed after first-line treatment and at least one second-line therapy including rituximab and/or TPO-RA.

DETAILED DESCRIPTION:
Primary immune thrombocytopenia is an autoimmune disease associated with a reduced peripheral blood platelet count. The first-line treatment is corticosteroids. Splenectomy, rituximab, and thrombopoietin receptor agonists (TPO RAs, such as Etrapopar and Romistine) are commonly used as second-line therapy. However, many of the treatments used achieve few lasting remissions. About 20% - 30% of patients have inadequate or no response to first-line and second-line treatment, and would develop into recurrent/refractory (r/r) ITP.

A branch of pathogenesis for ITP has been revealed that plasma cells secrete pathogenic antibodies directed against platelet and red blood cell antigens. Antiplatelet specific plasma cells have been detected in the spleen of patients with rituximab refractory ITP. In those refractory cases, persistent autoreactive long-lived plasma cells in the bone marrow could explain treatment failure.

Daratumumab, an anti-CD38 monoclonal antibody developed to target tumoral plasma cells in multiple myeloma, was recently found to be effective in antibody-mediated diseases, such as autoimmune cytopenia following hematopoietic stem cell transplantation, systemic lupus and also ITP.

This study will evaluate the safety and biologic activity of Daratumumab in r/r primary ITP who fail to respond to at least one previous second-line therapy. The study will enroll approximately 20 participants. This trial will be conducted in China. All participants will be followed for at least 16 weeks after the 8 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥18 years.
* Diagnosed with ITP that has persisted for ≥3 months and with a platelet count of <30 X 109/L measured within 2 days prior to inclusion.
* Failure to achieve response or relapse after corticosteroid therapy, and at least one second-line therapy including rituximab and/or TPO-RA.
* If receiving emergency care for ITP, treatment should be stopped >2 weeks before first dose.
* A positive result to the ELISA test to detect antibody against GPIIb/IIIa or GPIIb/IIIa and GPIb/IX within 1 week prior to inclusion.
* With normal hepatic and renal functions.
* ECOG Performance Status ≤ 2.

February 16, 2023 After approval by the Ethics Committee on , subjects no longer require platelet glycoprotein autoantibodies positivity upon enrollment.

Exclusion Criteria:

* Received any treatment of anti-CD38 antibody drug.
* Has been diagnosed with malignancy and/or liver failure, heart failure and renal failure.
* Known previous infection or seropositivity for HIV, Hepatitis B, Hepatitis C, Cytomegalovirus, EB virus, Syphilis.
* Any clinically overt hemorrhage.
* Has been diagnosed with cardiac disease, arrhythmia and/or severe or uncontrollable hypertension
* Known pulmonary embolism, thrombosis and/or atherosclerosis.
* Has been received allogeneic stem cell transplantation or organ transplantation.
* Patients with history of current or past psychiatric disease that might interfere with the ability to comply with the study protocol or give informed consent.
* Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-12-10 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate of response after daratumumab treatment | 8 weeks
  The proportion of patients with 2 consecutive platelet counts of ≥ 50×109/L within 8 weeks
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] of daratumumab | 24 weeks
  Incidence, severity, and relationship of treatment emergent adverse events after daratumumab treatment

SECONDARY OUTCOMES:
The proportion of patients with ≥2 consecutive platelet counts (separated by ≥7 days) of ≥30 × 109/L and a ≥2-fold increase from the baseline count within 8 weeks | 8 weeks
  The proportion of patients with ≥2 consecutive platelet counts (separated by ≥7 days) of ≥30 × 109/L and a ≥2-fold increase from the baseline count within 8 weeks.
Time to first platelet count of ≥50 × 109/L without salvage therapy. | 24 weeks
  Time to first platelet count of ≥50 × 109/L without salvage therapy.
Overall response rate at week 8 and week 24 | 24 weeks
  Complete response (CR) : 2 or more consecutive monitored platelet counts ≥100 × 109/L without bleeding symptoms,with an interval of at least 7 days; Partial response (PR) : 2 or more consecutive monitored platelet counts ≥30 × 109/L, at least a double baseline count (separated by ≥7 days), and no bleeding symptoms. Overall response (OR) : CR or PR.
Complete response rate at week 8 and week 24 | 24 weeks
  Complete response (CR) : 2 or more consecutive monitored platelet counts ≥100 × 109/L without bleeding symptoms,with an interval of at least 7 days.
Cumulative response duration of platelet count of ≥30 × 109/L and a platelet count doubling from the baseline within 24 weeks | 24 weeks
  Cumulative response duration of platelet count of ≥30 × 109/L and a platelet count doubling from the baseline within 24 weeks.
Durable sustained platelet count response rate | 24 weeks
  Durable sustained platelet count response rate is defined as the proportion of subjects with platelet counts of ≥30 × 109/L for at least six of the eight visits between weeks 17 and 24 of the study.
WHO bleeding score at baseline and at week 8 and 24 after treatment | 24 weeks
  WHO bleeding score at baseline and at week 8 and 24 after treatment. The WHO Bleeding Scale is a measure of bleeding severity with the following grades: grade 0 = no bleeding, grade 1= petechiae, grade 2= mild blood loss, grade 3 = gross blood loss, and grade 4 = debilitating blood loss.
The proportion of subjects with concomitant medication reduction or discontinuation | 24 weeks
  The proportion of subjects with concomitant medication reduction or discontinuation within 24 weeks.
The proportion of subjects receiving rescue medications | 24 weeks
  The proportion of subjects receiving rescue medications within 24 weeks.
Changes in immunoglobulin levels | 24 weeks
  Changes in immunoglobulin levels before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, M.D., Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Chinese Academy of Medical Science and Blood Disease Hospital, Tianjin, Tianjin Municipality, China